CLINICAL TRIAL: NCT00445185
Title: A Study to Evaluate the Persistence of Anti-HBs Antibodies at Months 12, 24 and 36 in Pre-dialysis or Dialysis Patients Who Have Received a Primary Vaccination Course of Either Henogen's HBV Vaccine, HB-AS02V or GSK Biological's Fendrix™
Brief Title: Study Evaluating Persistence of Anti-HBs Antibodies in Uraemic Patients Receiving Henogen's HBV Vaccine, or Fendrix™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henogen (Industry)
Responsible Party: Sophie Houard CSO, Henogen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HN015/HBV-EXT001
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Hepatitis B
Keywords: Dialysis; Pre-dialysis; Hepatitis B vaccine; vaccine
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Henogen Hepatitis B vaccine for uremic patients
  Interventions: Biological: Henogen HB vaccine
- 2 (Active Comparator): Fendrix hepatitis B vaccine for uremic patients
  Interventions: Biological: Fendrix vaccine

INTERVENTIONS:
Biological: Henogen HB vaccine — Month 12, 24 and 36
  Arms: 1
Biological: Fendrix vaccine — Month 12, 24 and 36
  Arms: 2

SUMMARY:
The current extension study will assess the persistence of anti-HBs antibodies at Months 12, 24 and 36 after primary vaccination with Henogen's HBV vaccine or Fendrix™. This protocol posting deals with the objectives & outcome measures of the extension phase at Months 12, 24 and 36. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT00291941).

DETAILED DESCRIPTION:
Subjects who received complete full vaccination with Henogen HBV adjuvanted vaccine or Fendrix™ will participate in this persistence study for three long-term time points (12, 24 and 36 months after the first dose of primary vaccination). Blood sampling will be done at each time point to measure immune persistence.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject/ from the parent/ guardian of the subject.
* Subjects who completed the full course of primary vaccination.

Exclusion Criteria:

* Immunosuppression caused by the administration of parenteral steroids or chemotherapy.
* Any confirmed or suspected human immunodeficiency virus (HIV) infection.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | Months 12, 24 and 36.

SECONDARY OUTCOMES:
Quality of immune response | Month 12, 24 and 36
SAEs retrospective reporting | Month 12, 24 and 36
RF-1 like antibody concentrations in the subset of subjects for whom this analysis was done at the primary study (HN014/HBV-001). | Month 12, 24 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Joëlle Nortier, MD, PhD, Principal Investigator — ULB Hôpital Erasme Département de Néphrologie
Locations (23):
- Belgium (13):
  - O.L.Vrouwziekenhuis Aalst, Aalst
  - RHMS La Madeleine ATH, Ath
  - RHMS Clinique Louis Caty Baudour, Baudour
  - CHU Brugmann (site V Horta) Service de néphrologie, Brussels
  - ULB Hôpital Erasme Département de Néphrologie, Brussels
  - AZ -VUB Dienst Nefrologie, Brussels
  - Cliniques universitaires Saint Luc, Brussels
  - CHU Hôpital civil de, Charleroi
  - UZ Gent, Ghent
  - CHU Tivoli, La Louvière
  - UZ Gasthuisberg Leuven Nierziekten, Leuven
  - CHU Andre VESALE, Montigny-le-Tilleul
  - RHMS TournayService de néphrologie, Tournai
- Czechia (5):
  - Hospital JihlavaVrchlického, Jihlava
  - Regional Hospital Liberec, Liberec
  - University Hospital with Outpatient Clinic Ostrava, Ostrava
  - Dept. of Internal Medicine StrahovSermirska 5, Prague
  - Masaryk´s Hospital Socialni pece 3316/12A, Ústí nad Labem
- Hungary (5):
  - St. Rókus Hospital, Budapest
  - St. István Hospital, Budapest
  - Petz Aladár Teaching Hospital, Győr
  - Pest County Flór Ferenc Hospital, Kistarcsa
  - Vas and Szombathely County Markusovszky Hospital, Szombathely

REFERENCES:
- [Derived] Surquin M, Tielemans C, Nortier J, Jadoul M, Peeters P, Ryba M, Roznovsky L, Doman J, Barthelemy X, Crasta PD, Messier M, Houard S. Anti-HBs antibody persistence following primary vaccination with an investigational AS02(v)-adjuvanted hepatitis B vaccine in patients with renal insufficiency. Hum Vaccin. 2011 Sep;7(9):913-8. doi: 10.4161/hv.7.9.16225. Epub 2011 Sep 1. PMID 21892006